CLINICAL TRIAL: NCT02699268
Title: Validation of VoluSense Pediatrics, a New Method of Infant Spirometry Based on Electromagnetic Inductance Plethysmography
Brief Title: A Clinical Study Aiming to Validate the Equipment: VoluSense Pediatrics (VSP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: REK Vest 2010/496-8
Record Dates: First submitted 2015-12-01; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Lung Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants (term borns and preterm borns): Intervention: simultaneous lung function measurement using VoluSense Pediatrics and a mask-based method with an ultrasonic flowmeter (EcoMedics Exhalyzer)
  Interventions: Other: Lung function measurement

INTERVENTIONS:
Other: Lung function measurement — The infants will be exposed to lung function measurements performed by a new metod (Volusense Pediatrics) and a validated method (EcoMedics Exhalyzer D). The two Methods will be compared. This is not an intervential study, but a study aiming to validate a New Method versus an old method

SUMMARY:
This is a cross-sectional observational study, aiming to validate the accuracy of tidal breathing measurements in infants made by VoluSense Pediatrics, a lung function method based on electromagnetic inductance plethysmography, compared to an ultrasonic flowmeter. VoluSense Pediatrics consists of a flexible vest placed around the torso of the baby, and changes in tidal volume and flow is measured. The study will enable a better understanding of the usefulness of this equipment. The equipment is made by VoluSense Norway AS, and is owned by Haukeland University Hospital.

DETAILED DESCRIPTION:
All infants will be assessed at the pediatric department at Haukeland University Hospital, and all data obtained by the same two investigators (Bentsen and Olsen). The infants will be dressed in the appropriate-sized vest selected according to the length from the armpit to the hip of the child. Care will be taken to ensure that the vest fits snugly around the torso and that the width of the copper wire zig-zag coveres the entire thorax and abdomen including the pubic region. The vest will be applied directly to the skin; neither body nor diaper will be worn underneath. The infants will then be fed before they will be placed supine in a cot and encouraged to sleep. No sedation will be used. Once the infant has fallen asleep, data will be collected with VSP for 2-3 minutes before the Exhalyzer D® neonatal facemask connected in series with the ultrasonic flow sensor will be placed gently, but firmly over the infant's mouth and nose, ensuring a good seal. Once the facemask is in place, a marker will be inserted in the VSP recording. The Exhalyzer D® measurement will be started about thirty seconds after the facemask has been put on, to allow adaptation to the facemask. Simultaneous recording using both devices will then be done for about 1 minute before the mask will be removed. New markers will be inserted in the VSP recording as the Exhalyzer D® measurement is started and stopped facilitating analysis of the same breathing cycles.

Data will be analysed and graphs will be created with SPSS version 22 (IBM SPSS Statistics, New York, US) and MedCalc version 13.1 (MedCalc Software, Mariakerke, Belgium). Bland-Altman plots will be used to visualize agreement between the two measurement techniques. For each pair of measurements, the pairwise mean of the breathing parameters will be plotted on the x-axis, and the pairwise difference expressed as a percentage of their mean value on the y-axis. The mean difference and the 95% limits of agreement and their confidence intervals will be represented by horizontal lines in the graphs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term born or preterm born babies ≥ 2000 grams.

Exclusion Criteria:

* Being in an unstable clinical condition.
* Weight < 2000 grams.

Ages: 2 Days to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term born and preterm born babies ≥ 2000 grams.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Tidal volume. Unit is milliliter | 1 hour
  Tidal volume will be measured using the two Methods and compared using Bland-Altman statistics

SECONDARY OUTCOMES:
Respiratory Rate. Unit is counts per minute | 1 hour
  Respiratory rate will be measured using the two Methods and compared using Bland-Altman statistics
Peak tidal expiratory flow (TPTEF). Unit is ml/sec | 1 hour
  TPTEF will be measured using the two Methods and compared using Bland-Altman statistics
the ratio of inspiratory to expiratory time (Ti/Te). This is a ratio, and thus no unit | 1 hour
  Ti/Te will be measured using the two Methods and compared using Bland-Altman statistics
The ratio of tidal expiratory flow at 50% of expired volume to peak tidal expiratory flow (TEF 50/PTEF). | 1 hour
  TEF 50/PTEF will be measured using the two Methods and compared using Bland-Altman statistics
Total expiratory time (Tptef/Te). This is a ratio, and thus no unit | 1 hour
  Tptef/Te will be measured using the two Methods and compared using Bland-Altman statistics

CONTACTS AND LOCATIONS:
Overall Officials: Trond Markestad, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Pediatric department, NICU, Bergen, Western Norway, Norway

IPD SHARING:
Plan to Share IPD: No